CLINICAL TRIAL: NCT03874091
Title: Clinical Effectiveness of Erector Spinae Plane Block in Peri-operative Analgesia for Laparoscopic Kidney Procedures
Brief Title: Clinical Effectiveness of Erector Spinae Plane Block in Peri-operative Analgesia for Laparoscopic Nephrectomy/Nephron Sparing Surgery (NSS)/Hynes-Anderson Procedures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MedUnivLapESPblock
Record Dates: First submitted 2019-01-21; First posted 2019-03-14 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2020-03

CONDITIONS: Erector Spinae Plane Block
Keywords: Erector Spinae Plane block; ESP block; Laparoscopic Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA group (Active Comparator): Patients will receive general anaesthesia for laparoscopic nephrectomy/NSS/ Hynes Anderson procedures. Analgesia will be provided by titration of fentanyl during surgery. An intravenous patient controlled morphine pump will be used postoperatively.
  Interventions: Drug: Morphine PCA pump
- ESP group (Experimental): Patients will receive general anaesthesia with bilateral ESP block for laparoscopic nephrectomy/NSS/ Hynes Anderson procedures. Catheter will be inserted in the erector spinae plane on the side of surgery. Postoperatively patients will get continuous infusion of 0,125% Bupivacaine+Adrenaline to the catheter for 24h and PCA morphine pump intravenously.
  Interventions: Procedure: bilateral ESP block with 0,25% Bupivacaine+ Adrenaline; Procedure: ESP block continuous infusion with 0,125% Bupivacaine+Adrenaline; Drug: Morphine PCA pump

INTERVENTIONS:
Procedure: bilateral ESP block with 0,25% Bupivacaine+ Adrenaline — Regional anaesthesia technique performed under ultrasound guidance before surgery
  Arms: ESP group
Procedure: ESP block continuous infusion with 0,125% Bupivacaine+Adrenaline — Continous infusion of Local Anaesthetic (LA) given postoperatively via the catheter.
  Arms: ESP group
Drug: Morphine PCA pump — Morphine given postoperatively.

SUMMARY:
62 patients age of 20 to 85, (ASA) physical status I-III undergoing laparoscopic nephrectomy/NSS/Hynes Anderson procedures in 1st Department of Anesthesiology in Warsaw will be enrolled in the study. Patients will be randomised into 2 groups - patients from the first group will undergo General Anaesthesia (GA) with intravenous analgesia peri-operatively, patients from the second group will receive GA plus the Erector Spinae Plane Block (ESP block) bilaterally performed under ultrasound guidance with catheter left on the side of surgery. Ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the Th7 spinous process. Three muscles will be identified superficial to the hyperechogenic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. An 8-cm 18-gauge block needle will be inserted in a cephalad-to-caudad direction until the tip gets in the interfascial plane between rhomboid major and erector spinae muscles, as evidenced by visualization of local anesthetic spreading in a linear pattern between erector spinae and the bony acoustic shadows of the transverse processes. . Patients in this group will be anesthetized with 20ml 0,25% bupivacaine + Adrenaline 1:200 000 for each side. ESP block will be performed at the level of Th7-8 after proper positioning he patient in the sitting position before GA then standard technique of catheter application will be applied. After the surgery the elastomeric pump will be attached to the catheter with 0,125% bupivacaine with Adrenaline 1:200 000. Anaesthesia will be standardised In the both groups.

ELIGIBILITY:
Inclusion Criteria:

* pts undergoing laparoscopic nephrectomy/NSS/Hynes Anderson procedures in 1st Department of Anaesthesiology in Warsaw
* pts consented for the study prior to surgery
* ASA 1-3

Exclusion Criteria:

* Pts without consent for trial
* Pts ASA 4-5
* Coagulation abnormalities
* Allergy to local anesthetics
* Skin lesions in the place of needle insertion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Morphine Requirements | 24 hours post surgery
  Patient Controlled Analgesia (PCA) morphine consumption in both groups will be recorded.

SECONDARY OUTCOMES:
Intraoperative Fentanyl Requirements | Time of surgery.
  Fentanyl consumption in both groups will be recorded

OTHER OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | 24 hours post surgery.
  Postoperative nausea and vomiting will be recorded if occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Warsaw University Center, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No